CLINICAL TRIAL: NCT06198959
Title: Heat Loss in Humans Covered With Full-Body Blankets Connected to Different Warming Devices
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: The Surgical Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 22-871
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Heat Transfer by Clinical Warming Devices

STUDY DESIGN:
Intervention Model Description: The investigators propose a single-center multiple crossover randomized trial to determine cutaneous heat transfer with four warming devices and five blankets. Cutaneous heat loss/ gain will be measured with thermal flux transducers in unanesthetized volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- ABCDE (Experimental): A. Volunteers will be covered with the Adult Blanket plus, MA2220 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes. B. After a 40 minutes washout period, the volunteers will be covered with the Premium Adult Blanket, 3320 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes. C. After a 40-minute washout period, the volunteers will be covered with the Blanket full body, 30000 connected to the 3M, Bair Hugger, Blower 775 for 30 minutes. D. After a 40-minute washout period, the volunteers will be covered with the FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system for 30 minutes. E. Finally and after a last 40-minute washout period, the volunteers will be covered with the Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system for 30 minutes.
  Interventions: Device: Adult blanket plus, MA2220 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Premium adult blanket, 3320 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775; Device: FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system.; Device: Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system
- BDECA (Experimental): B. Volunteers will be covered with the Premium Adult Blanket, 3320 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes. D. After a 40-minute washout period, the volunteers will be covered with the FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system for 30 minutes. E. After a 40-minute washout period, the volunteers will be covered with the Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system for 30 minutes. C. After a 40-minute washout period, the volunteer will be covered with the Blanket full body, 30000 connected to the 3M, Bair Hugger, Blower 775 for 30 minutes. A. Finally and after a last 40-minute washout period, the volunteers will be covered with the Adult Blanket plus, MA2220 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes.
  Interventions: Device: Adult blanket plus, MA2220 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Premium adult blanket, 3320 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775; Device: FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system.; Device: Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system
- CEBAD (Experimental): C. Volunteers will be covered with the blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775 for 30 minutes. E. After a 40-minute washout period, the volunteers will be covered with the Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system for 30 minutes. B. After a 40-minute washout period, the volunteers will be covered with the Premium Adult Blanket, 3320 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes. A. After a 40-minute washout period, the volunteers will be covered with the adult blanket plus, MA2220 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes. D. Finally and after a last 40-minute washout period, the volunteers will be covered with the FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system for 30 minutes.
  Interventions: Device: Adult blanket plus, MA2220 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Premium adult blanket, 3320 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775; Device: FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system.; Device: Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system
- DCAEB (Experimental): D. Volunteers will be covered with the FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system for 30 minutes. C. After a 40-minute washout period, the volunteers will be covered with the blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775 for 30 minutes. A. After a 40-minute washout period, the volunteers will be covered with the adult blanket plus, MA2220 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes. E. After a 40-minute washout period, the volunteers will be covered with the blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system for 30 minutes. B. Finally and after a last 40-minute washout period, the volunteers will be covered with the Premium Adult Blanket, 3320 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes.
  Interventions: Device: Adult blanket plus, MA2220 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Premium adult blanket, 3320 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775; Device: FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system.; Device: Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system
- EADBC (Experimental): E. Volunteers will be covered with the blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system for 30 minutes. A. After a 40-minute washout period, the volunteers will be covered with the adult blanket plus, MA2220 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes. D. After a 40-minute washout period, the volunteers will be covered with the FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system for 30 minutes. B. Finally and after a last 40-minute washout period, the volunteers will be covered with the Premium Adult Blanket, 3320 connected to the Mistral Air, Blower MA1200-PM system for 30 minutes. C. Finally and after a last 40-minute washout period, the volunteers will be covered with the blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775 for 30 minutes.
  Interventions: Device: Adult blanket plus, MA2220 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Premium adult blanket, 3320 blanket connected to the Mistral Air, Blower MA1200-PM system.; Device: Blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775; Device: FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system.; Device: Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system

INTERVENTIONS:
Device: Adult blanket plus, MA2220 blanket connected to the Mistral Air, Blower MA1200-PM system. — Evaluate cutaneous heat loss/ gain using thermal flux transducers while volunteers are covered with the Adult Blanket plus, MA2220 blanket connected to the Mistral Air, Blower. MA1200-PM system for 30 minutes.
Device: Premium adult blanket, 3320 blanket connected to the Mistral Air, Blower MA1200-PM system. — Evaluate cutaneous heat loss/ gain using thermal flux transducers while volunteers are covered with the premium adult blanket, 3320 blanket connected to the Mistral Air, Blower MA1200-PM system.
Device: Blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775 — Evaluate cutaneous heat loss/ gain using thermal flux transducers while volunteers are covered with the blanket full body, 30000 blanket connected to the 3M, Bair Hugger, Blower 775 system.
Device: FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system. — Evaluate cutaneous heat loss/ gain using thermal flux transducers while volunteers are covered with the FilteredFlo® Air Blanket connected to the WarmAir® Convective Warming system.
Device: Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system — Evaluate cutaneous heat loss/ gain using thermal flux transducers while volunteers are covered with the Blanket Full Body blanket (CLM0101) connected to the Care Essential, Cocoon, Blower CWS5000 system.

SUMMARY:
The investigators propose a single-center multiple crossover randomized trial to determine the efficacy of four warming devices and five warming blankets. The investigators will measure cutaneous heat loss/ gain using thermal flux transducers in unanesthetized volunteers.

DETAILED DESCRIPTION:
The investigators propose a single-center, assessor-Blinded, multiple crossover randomized trial to determine the efficacy of four warming devices and five blankets. The investigators will measure cutaneous heat loss/ gain using thermal flux transducers in unanesthetized volunteers.

American Society of Anesthesiologists (ASA) physical status 1 and 2 adults with body-mass index 20-33 kg/m2 will be included in this study. Volunteers will be excluded if they have serious skin lesions, history of allergy or skin sensitivity to tape or adhesive materials, serious vascular disease in the arms including Raynaud's Syndrome, or a history of recent fever or infection.

20 volunteers will be randomized to one of 5 different sequence groups: 1. Mistral Air, Blower MA1200-PM. plus the Adult Blanket plus, MA2220, 2. Mistral Air, Blower MA1200-PM plus the Premium Adult Blanket, 3320, 3. 3M, Bair Hugger, Blower 775 plus Blanket full body, 30000, 4. Smiths Medical, Blower L1-CW-100V, plus Blanket full body SWU-2001, 5. Care Essential, Cocoon, Blower CWS5000 plus Blanket Full Body blanket (CLM0101).

ELIGIBILITY:
Inclusion Criteria:

* Body-mass index 20-33 kg/m2
* Age 18-40 yrs.
* ASA Physical Status 1-2.

Exclusion Criteria:

* Serious skin lesions
* History of allergy or skin sensitivity to tape or adhesive materials
* History of serious vascular disease in the arms, including Raynaud's Syndrome
* History of recent fever or infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Heat transfer, thermal flux | 30 minutes
  While using one of the 5 different warming blanket and warming blower systems, heat transfer will be measured on at 15 sites: Head, upper arm, forearm, hand, finger, back, chest, abdomen, medial thigh, lateral thigh, posterior thigh, anterior calve, posterior calves, foot and toe.

SECONDARY OUTCOMES:
Thermal comfort | 30 minutes
  After completing 30 minutes using the warming system, before removing the warming blanket, volunteers will rate their thermal comfort in a 0-100 mm scale. the minimum is 0 representing the coldest and the maximum value is 100 mm representing the hotest sensation the participant can report.

CONTACTS AND LOCATIONS:
Overall Officials: sessled@ccf.org Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States